CLINICAL TRIAL: NCT05894083
Title: A Phase II Study for p16+ Oropharyngeal Cancer PerSonalized De-escalation Treatment at University of MIchigan (CuSToMIze)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2022.043; HUM00221848 (Other: University of Michigan)
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Oropharyngeal Cancer; Squamous Cell Carcinoma of the Oropharynx
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Surgical Procedures, Operative; Chemoradiotherapy; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator): Surgery followed by risk-adjusted adjuvant treatment (observation, radiation, or chemoradiation).
  Interventions: Procedure: Surgery; Combination Product: Chemoradiation; Other: Observation; Radiation: Post-operative radiation
- Definitive CRT (Experimental): Risk-adjusted definitive chemoradiation.
  Interventions: Combination Product: Chemoradiation

INTERVENTIONS:
Procedure: Surgery — Cohort A will undergo initial surgical resection of the primary and neck dissection with pathologic features directing predetermined adjuvant treatment. Pathology of the primary and nodal specimens will then be reviewed as to determine the next intervention per protocol. Based on operative findings including degree of nodal involvement, extracapsular spread, perineural invasion, and lymphovascular involvement, patients will be designated to adjuvant treatment arms consisting of observation, adjuvant radiation, or adjuvant chemoradiation.
  Arms: Surgery
Combination Product: Chemoradiation — Patients will receive an initial plan with a single prescription of 30 Gy in 15 fractions to PTV_High and PTV_Low with RT given once daily, 5 days a week (Monday through Friday). After analysis of mid-treatment PET/CT, the remaining radiation treatment will be delivered as a conedown to the gross disease only. Patients will be planned to receive a total dose of 70 Gy, 54 Gy, or 44 Gy to PTV_High in 2 Gy per fraction.
Other: Observation — Cohort A will undergo initial surgical resection of the primary and neck dissection with pathologic features directing predetermined adjuvant treatment. Pathology of the primary and nodal specimens will then be reviewed as to determine the next intervention per protocol. Based on operative findings including degree of nodal involvement, extracapsular spread, perineural invasion, and lymphovascular involvement, patients will be designated to adjuvant treatment arms consisting of observation, adjuvant radiation, or adjuvant chemoradiation.
  Arms: Surgery
Radiation: Post-operative radiation — Patients will receive adjuvant radiation based on pathologic features.Total radiation treatment doses and prescriptions will include 36 Gy in 18 fractions, 50 Gy in 25 fractions and 60 Gy in 30 fractions.
  Arms: Surgery

SUMMARY:
Single center, non-randomized Phase II study enrolling Stage I-II p16+ oropharyngeal cancer patients to one of two de-escalation treatment paradigms: (1) receive surgery followed by observation or risk-adjusted adjuvant radiation (+/-chemo), or (2) individualized adaptive definitive chemoradiation (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have FDG-avid (maximum SUV ≥ 4.0) (from PET scan of any date, any scanner) and histologically or cytologically proven squamous cell carcinoma of the oropharynx (tonsil, base of tongue, oropharyngeal wall, soft palate) or unknown primary that is p16 positive by immunohistochemistry or HPV positive by in situ hybridization
* Clinical stage: Stage I-II AJCC 8th edition staging
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

  * History/physical examination, including documentation of weight within 4 weeks prior to registration;
  * For Cohort B, FDG-PET/CT scan for staging within 6 weeks prior to registration. For Cohort A, acceptable imaging for staging can include diagnostic CT neck/chest or PET-CT within 6 weeks prior to registration
  * Zubrod Performance Status 0-1 within 4 weeks prior to registration;
  * Age ≥ 18;
  * Able to tolerate PET/CT imaging required to be performed
* For Cohort A, tumors must be potentially surgically resectable via a transoral approach, at the discretion of the treating surgeon. Additionally, they must have 0-2 clinically positive LNs on diagnostic CT or PET-CT according clinical consensus of the treatment team
* For both cohorts, CBC required within 4 weeks prior to registration. For Cohort B, CBC/differential obtained within 4 weeks prior to registration on study, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3;
  * Platelets ≥ 100,000 cells/mm3;
  * Hemoglobin ≥ 8.0 g/dL
* Serum creatinine within normal institutional limits or a creatinine clearance ≥ 45 ml/min within 4 weeks prior to registration.
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study.
* The patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* cT4, cN3, or cM1 disease (also explained as AJCC 8th edition clinical staging,)
* Patients with radiographic ECE or matted lymph nodes, defined as three nodes abutting one another with loss of intervening fat plane that is a replaced with radiologic evidence of extracapsular spread.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible);
* Any prior therapy for the study cancer; note that prior chemotherapy for a different cancer is allowable if >3 years prior to study;
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
* Prior allergic reaction or hypersensitivity reactions to paclitaxel, carboplatin or other platinum containing products. This also includes patients with a history of severe hypersensitivity reaction to products containing Cremophor EL.
* Severe, active co-morbidity, defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;

  * Transmural myocardial infarction within the last 3 months;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic Obstructive Pulmonary Disease (COPD) exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition. Note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
  * Severe bone marrow depression or significant bleeding
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* For Cohort B, poorly controlled diabetes (defined as fasting glucose level > 200 mg/dL) despite 2 attempts to improve glucose control by fasting duration and adjustment of medications. Patients with diabetes will preferably be scheduled in the morning and instructions for fasting and use of medications will be provided in consultation with the patients' primary physicians.
* Active enrollment on another clinical trial involving active treatment for the study cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Loco-regional recurrence free survival (LR-RFS) rate | 2 years
  LR-RFS is defined as the difference between the date of the first treatment to the date of the first of the following events: death (any cause) or loco-regional progression. LR-RFS rates will be reported using Kaplan Meier (KM) estimates at 2 years.

SECONDARY OUTCOMES:
Progression free survival (PFS) rate | 2 years
  PFS is defined as the difference between the date of the first therapy to the date of the first of the following events: death (any cause) or disease progression (local, regional, distant, defined as per section 7.1). PFS data will be censored on the date of the last tumor assessment on study for subjects who do not have objective tumor progression and who do not die while on study.
Disease specific survival (DSS) rate | 2 years
  DSS is defined as the difference between the date of the first treatment intake to the date of death due to oropharyngeal cancer.
Overall survival (OS) rate | 2 years
  OS is defined as the difference between the date of the first treatment intake to the date of death (any cause).
Patterns of failure (locoregional relapse versus distant) | 2 years
  Defined as the proportion of patients who progressed in any location and whether the first progression was local, regional or distant or in multiple locations.
Acute toxicity | up to 3 months post definitive treatment completion {section 2.4.2 of protocol states only 3 months but 2.2 states 3 and 6 months - will clarify with study team}
  Defined as the proportion of patients with available toxicity data and the proportion of all treated patients through cumulative incidence estimates with death treated as a competing risk and censoring for patients lost to follow-up (FU).
Late toxicity | up to 24 months post definitive treatment completion
  Defined as the proportion of patients with available toxicity data and the proportion of all treated patients through cumulative incidence estimates with death treated as a competing risk and censoring for patients lost to follow-up (FU).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Mierzwa, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided